CLINICAL TRIAL: NCT06204003
Title: Naturally Produced Cannabinoids for Pain Management and Neuroprotection From Concussion During Participation in Contact Sports: Dose Escalation
Brief Title: Cannabinoids for Pain Management and Neuroprotection From Concussion
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Regina (Other)
Collaborators: National Football League (NFL) (Unknown); My Next Health Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3455; NFL-CBD-01 (Other: URegina)
Record Dates: First submitted 2023-07-24; First posted 2024-01-12 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: All participants will receive placebo at Day 0. CBD 5 mg/kg will begin Day 15. CBD 10 mg/kg will begin Day 30. CBD 15 mg/kg will begin Day 45. CBD 20 mg/kg will begin Day 60. CBD 25 mg/kg will begin Day75. CBD 30 mg/kg will begin Day 90.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): When participants start the CBD, they will be started on a low dose of CBD, beginning at 5 mg CBD/kg body mass, and then increased by 5 mg/kg every 2-weeks until 30 mg CBD/kg body mass is taken.
  Interventions: Drug: Cannabis/Hemp Isolate Extract

INTERVENTIONS:
Drug: Cannabis/Hemp Isolate Extract — Formulation: CBD (99%; 0.1% THC isolate)
  Other Names: Herbal Extract with a high CBD

SUMMARY:
The goal of this open-label, placebo-controlled, dosage escalation study is to learn about the safety of a Cannabis/Hemp Isolate Extract in normal healthy adults engaged in elite contact sport competition.

The main question it aims to answer is:

• Are cannabis/hemp-based products with high CBD safe, well-tolerated and without adverse physiological and psychological dysfunction, when administered on a daily basis?

Participants will:

* be given CBD and a placebo. The placebo will be taken for 2 weeks prior to starting the CBD. Participants will start on a low dose of CBD, beginning at 5 mg CBD/kg body mass, which will be increased by 5 mg/kg every 2-weeks until 30 mg CBD/kg body mass is taken;
* have blood samples taken to analyse how much CBD is used in the body and for how long it lasts in the body (pharmacokinetics and pharmacodynamics);
* have saliva samples collected for genetic analysis;
* undergo testing sessions, which will include psychological and health questionnaires, equipment to record signals from the brain and heart, and safety laboratory tests.

DETAILED DESCRIPTION:
This research project will be a Phase I clinical trial to test the safety, efficacy and tolerability of the drug formulation. Specifically, the investigators will use a dose escalation study with all participants taking a placebo before starting the CBD regimen. This study is designed to investigate anti-inflammatory and neuroprotection of the CBD formulation to determine whether it can be used on a daily basis safely during the periods of intensive exercise (resistance) training during the off-season prior to competition.

The primary research hypothesis is that cannabis/hemp-based products with high CBD are safe, well-tolerated and do not cause adverse physiological and psychological dysfunction when administered on a daily basis. Specifically, the investigators will investigate the pharmacokinetic, physiological, and psychological effects of CBD. The investigators hypothesize that the CBD formulations will be non-intoxicating (non-psychotropic), safe, well-tolerated and do not cause adverse physiological or psychological dysfunction.

Secondary research hypotheses for this clinical trial:

1. Pharmacokinetic data will provide the investigators with the 'optimal' formulation for daily administration for neuroprotection from concussion
2. Plasma levels of CBD and/or its active metabolites will correlate with cerebrovascular, neurophysiology and cardiovascular physiology outcome variables.
3. Saliva levels of CBD and/or its active metabolites will correlate with plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male adults between 18-35 years of age that compete in contact sport athletics
* No known cerebrovascular or cardiovascular complications
* Not habitual recreational users of cannabis (i.e., <1 day/week) or tobacco users
* Agree not to consume any other cannabis or tobacco products while enrolled in the study
* Agree to list any prescription medications being taken
* Ability to maintain commitment to all proposed biopsychological and health questionnaires, and neuro-physiological, physiological, perceptual-cognitive, and functional motor skills laboratory tests

Exclusion Criteria:

* Female
* Requirement to travel to the USA during study period; USA laws do not permit cross border with cannabis products
* Use of cannabis-based therapy within 2 months (participants who have previously used a cannabis based therapy may be included if they have a 2 month period without use of cannabis based therapy prior to enrolment in the study)
* Any level of cannabis in blood samples when sampled at the commencement of the study
* Medically supervised for anxiety, depression, or other neurological conditions
* Initiation or dosage change of oral or injected steroids within past 3 months
* Allergy or known intolerance to any of the compounds within the study preparation
* Inability to attend assessments on a regular basis at the pre-determined times, or failure to take drug on a daily basis
* Clinically significant cardiac, renal or hepatic disease (as assessed by the site investigator)
* Concussion

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in cerebrovascular and cardiovascular physiology | Every 15 days from Day 0 to Day 104
  Monitor the participant's cerebrovascular and cardiovascular physiology before and after the dosage regimen
Incidence of potential harmful side effects | Every 15 days from Day 0 to Day 104
  Follow the participants enrolled in these studies at set intervals to monitor for potential harmful side effects of the high CBD cannabis/hemp extract. This will include bloodwork to assess for possible hematopoietic, renal or hepatic dysfunction, and pharmacokinetic and pharmacodynamic analysis of the dose escalation protocol

SECONDARY OUTCOMES:
Assessment of GABAergic activity | Every 15 days from Day 0 to Day 104
  Assess the inhibitory neurotransmitter δ-aminobutyric acid (GABAergic activity)
Change in pain intensity | Every 15 days from Day 0 to Day 104
  Pain Behaviour Measurement system (PBM) scale
Cerebral blood flow (transcranial Doppler) | Every 15 days from Day 0 to Day 104
  Assessment of cerebral hemodynamic activity
Cerebral oxygenation (near infrared spectroscopy) | Every 15 days from Day 0 to Day 104
  Assessment of cerebral hemodynamic activity
Change in QoL | up to day 104
  Assess quality of life (QOL) in study participants by scores on health questionnaires and medication use
Incidence of AEs | Through study completion, From Day 0 to Day 104
  Assess adverse events (AEs) in study participants by looking at sleepiness/lethargy, irritability, nausea/vomiting and diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Neary, Study Director — University of Regina; Payam Dehghani,, Principal Investigator — Saskatchewan Health Authority - Regina Area
Locations (2):
- Canada (2):
  - University of Regina, Regina, Saskatchewan
  - Pasqua Hospital, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neary JP, Singh J, Alcorn J, Laprairie RB, Dehghani P, Mang CS, Bjornson BH, Hadjistavropoulos T, Bardutz HA, Bhagaloo L, Walsh Z, Szafron M, Dorsch KD, Thompson ES. Pharmacological and physiological effects of cannabidiol: a dose escalation, placebo washout study protocol. BMC Neurol. 2024 Sep 12;24(1):340. doi: 10.1186/s12883-024-03847-1. PMID 39266961